CLINICAL TRIAL: NCT04194606
Title: CORRECT RADIAL RCT: CORonaRy Angiography and intErventions Via Distal vs Proximal aCcess - a Randomized Trial of Different Radial Puncture Sites
Brief Title: CORonaRy Angiography and intErventions Via Distal vs Proximal aCcess
Acronym: CORRECT Radial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. med. Karsten Schenke (Other)
Collaborators: Asklepios proresearch (Industry)
Responsible Party: Sponsor-Investigator, Dr. med. Karsten Schenke, Oberarzt - Consultant, Asklepios Kliniken Hamburg GmbH
Organization: Asklepios Kliniken Hamburg GmbH (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CORRECT Radial RCT 2019
Record Dates: First submitted 2019-12-07; First posted 2019-12-11 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Coronary Angiography; Coronary Artery Disease
Keywords: Anatomical snuffbox; Percutaneous coronary intervention; Radial access; Distal radial access; Radial artery occlusion; Coronary catheterization; Radial artery
MeSH Terms: conditions — Coronary Artery Disease; Arterial Occlusive Diseases | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, open Label randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Forearm radial access (Active Comparator): Patients who undergo coronary angiography or intervention by forearm radial artery access
  Interventions: Procedure: Use of radial artery for access for a coronary angiography or intervention
- Distal radial access (Experimental): Patients who undergo coronary angiography or intervention by accessing the distal radial artery in the area of the anatomical snuff-box
  Interventions: Procedure: Use of radial artery for access for a coronary angiography or intervention

INTERVENTIONS:
Procedure: Use of radial artery for access for a coronary angiography or intervention — After puncture of the radial artery in either the area of the anatomical snuffbox or the lower forearm following modified Seldinger technique a sheath will be advanced and a CAG or PCI will be performed. After the procedure is finished the sheath will be withdrawn and a standard closure device will be applied to achieve hemostasis. The choice of the patients side, the sheath, the catheters and the closing device will be at the discretion of the interventionalist.

SUMMARY:
The objective of the study is to determine that a coronary angiography (CAG) or percutaneous coronary intervention (PCI) via a distal puncture of the radial artery (distal transradial access, dTRA) leads to a lower rate of radial artery occlusion (RAO) while also showing that it has a similar success rate when compared to the traditional proximal (proximal transradial access, pTRA) puncture site.

DETAILED DESCRIPTION:
Cardiac catheterization is one of the most common invasive procedures worldwide. After demonstrating the superiority of the radial access over the femoral arterial approach, the radial artery puncture has become the first choice for elective and emergency coronary interventions. In addition to the often chosen access on the inside of the forearm, the course of the radial artery also allows a puncture further distal on the back of the hand. In the anatomical snuffbox, the diameter is still sufficient for the introduction of the usual sheath, however, the thrombogenic puncture at the proximal radial segment is avoided and a hemostasis by compression over the scaphoid is simplified.

This study is a prospective, open-label, randomized, multicenter study to systematically compare primary success rates and potential complications after distal transradial coronary angiography or coronary intervention versus proximal radial artery puncture over the wrist. Both puncture routes are well established in clinical routine and are used in both elective and emergency cardiac catheterization in the centers involved and worldwide. Systematic comparisons exist so far only in small series, but randomized and prospective data would be urgently needed in the frequent application. Both puncture sites are only 4-8 cm apart, so that many risks of a transradial examination (vascular injury and / or closure, perforation, spasm) are in principle common to both access sites.

The purpose of this study is to demonstrate the potential benefits of radial artery puncture in the back of the hand due to a reduced rate of chronic vascular occlusion compared to over the wrist, as well as complications (bleeding or nerve damage) and subjective tolerability ( Pain) systematically.

ELIGIBILITY:
Inclusion Criteria:

* Written consent to participate in the study
* Age ≥ 18 years
* Indication for coronary angiography or coronary intervention
* Palpable pulse of the proximal and distal radial artery on one or both arms

Exclusion Criteria:

* Hemodynamic instability (according to the criteria of cardiogenic shock: Hf> 120 / min and RR syst <90 mmHg)
* Intubated patients
* Sonographic evidence of occlusion of both radial arteries
* Pregnant or lactating women
* Patients that are currently or have within the last 30 days participated in a clinical trial
* Primarily planned bilateral radial access; e.g. in the context of a CTO recanalization
* Patients who are in a dependency / employment/ relationship with the study doctor or center
* Patients with bilateral hand or arm misalignment / paresis that makes a radial Access impossible
* Patients who do not speak German or who are unable to understand the nature, significance or scope of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2020-01-14 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Lower rate of forearm radial artery occlusion (RAO) | 30 days
  Use of color doppler ultrasound to assess the patency of the radial artery used in the index procedure.

SECONDARY OUTCOMES:
Puncture success rate of the randomized puncture site | During the procedure
  Comparison of the rate of successful Insertion of the sheath in each group
Access cross over rate | During the procedure
  Comparison of the rate of access site cross over in each group to complete the planned procedure
Duration of puncture | During the procedure
  Exact measurement of the duration of the puncture in seconds
Hematoma, bleeding and other complications | 48 hours
  Registration of complications associated with the procedure, hematoma size, bleeding according to the BARC Score
Use of standard questionaire to assess pain | 30 days
  Visual analog scale is used to assess pain
Incidence of vasospasm | during the procedure
  The incidence of vasospasm that necessitates additional medication or Forces Access site cross over is registered
Use of standard questionaire to assess Hand function | 30 days
  QuickDASH questionaire is used to assess Hand function

CONTACTS AND LOCATIONS:
Overall Officials: Karsten Schenke, MD, Principal Investigator — Asklepios Klinik Bambek Hamburg
Locations (3):
- Germany (3):
  - Klinikum Landkreis Erding, Erding, Bavaria
  - Sana Kliniken Düsseldorf GmbH, Düsseldorf, North Rhine-Westphalia
  - Asklepios Klinik Barmbek, Hamburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schenke K, Prog R, Joghetaei N, Sood N, Viertel A, Matthiesen T, Bott-Flugel L, Ohm S, Dill T, Gronefeld G. CORRECT RADIAL RCT. CORonaRy angiography and intErventions via distal vs proximal transradial aCcess-a randomized Trial of different RADIAL puncture sites. Clin Res Cardiol. 2026 Jan;115(1):99-111. doi: 10.1007/s00392-025-02759-5. Epub 2025 Nov 24. PMID 41284047